CLINICAL TRIAL: NCT05662124
Title: Comparison of Health Outcomes in a Remote Monitoring Programme Versus Usual Care in Interstitial Lung Disease
Brief Title: ILD: Health Outcomes in Remote Digital Monitoring Versus Usual Care
Acronym: REMOTE-ILD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: patientMpower Ltd. (Industry); Imperial College London (Other); University College, London (Other); Action for Pulmonary Fibrosis (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21SM6951
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Monitoring (Experimental): Patients in this arm will be asked to record their spirometry and oximetry three times weekly. This will be performed using a spirometer and oximeter which upload the results via bluetooth to the patientMpower app on their smartphones/tablets. These results are immediately available for review by their clinical teams who will be asked to review them at least once a fortnight.
  All patients will be asked to complete surveys at baseline, 3, 6, and 12 months and for clinical outcome data during the observation period to be collected.
  Interventions: Other: Remote monitoring
- Usual Care (No Intervention): Patients in this arm will undergo usual clinical care as planned by their medical team. They will be asked to complete surveys at baseline, 3,6 and 12 months and for clinical outcome data during the observation period to be collected.

INTERVENTIONS:
Other: Remote monitoring — Patients will download the patientMpower app and be provided with a spirometer (Spirobank Smart, MIR) and oximeter (Nonin) to record their spirometry and pulse oximetry which will upload to the application via Bluetooth for clinical review.
  Patients will be asked to upload measurements three times per week.
  Other Names: patientMpower app
  Arms: Remote Monitoring

SUMMARY:
Interstitial lung disease (ILD) is a collective term for a group of diseases where the lungs become scarred causing breathlessness.

This research project will assess if remote digital monitoring of frequent spirometry and pulse oximetry can provide an additional way to monitor ILD and provide information to support virtual consultations. Outcomes in the remote monitoring group will be compared with usual care alone over 12 months.

Patients taking part will be randomly allocated to remote digital monitoring or to usual care (with an equal chance of either). Remote monitoring will be performed using an app provided by patientMpower Ltd which patients will be able to download onto a smartphone or tablet. The study team will provide a spirometer and oximeter for patients to measure their lung function (spirometry) and oxygen saturations. These devices link to the app via Bluetooth to record all measurements. Patients will be asked to do these measurements three times a week. Clinical teams will be asked to review all measurements at least once a fortnight.

Health outcomes will be described and compared between the two groups.

DETAILED DESCRIPTION:
This study hopes to understand more about how remote digital monitoring of spirometry and pulse oximetry fits within the clinical care of patients with interstitial lung disease. This study will randomise patients to either remote monitoring or usual care and then collect information about the trajectory of their interstitial lung disease treatment and monitoring for the next 12 months to understand the impact of remote monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibrotic interstitial lung disease
* Aged at least 18 years
* Owns a smartphone or tablet device
* Has a mobile telephone number, email address and access to the internet at home
* In clinic lung function assessment within 6 months prior to study entry including spirometry and gas transfer measurement
* Intention to have at least two outpatient clinical reviews (either in person or virtual) within the study observation period of 12 months
* Willing to allow home monitoring of their health including spirometry and pulse oximetry data
* Understands how to use mobile technology (eg. has downloaded and used other "apps" on their mobile device; uses email)
* Demonstrates willingness to measure spirometry and pulse oximetry three times weekly for the duration of the observation period
* Fluent in English language
* Written or electronic informed consent

Exclusion Criteria:

* Unable to fulfil all inclusion criteria
* Cognitive impairment
* History of difficulties performing spirometry at previous clinic testing
* Contraindications to spirometry (for example previous pneumothorax, unstable cardiac status, known aortic or cerebral aneurysm)
* Serious concomitant conditions which place the patient at high risk of respiratory distress making them unsuitable to be managed at home.
* Current or recent (within the last 6 weeks before baseline) participation in another research project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Spirometry availability at clinical review at first and last clinic appointments during the study observation period | 12 months
  Number of patients who have spirometry recorded with the preceding 2 weeks for review at the first and last clinical reviews during the observation period

SECONDARY OUTCOMES:
Number of clinical reviews per patient | 12 months
  Average for each study arm
Proportion of clinical reviews which are virtual | 12 months
  Average for each study arm
Number of in-clinic lung function appointments per patient | 12 months
  Total number for each study arm
Number of patients who have chest CT scans | 12 months
  Total number for each study arm
Change in forced vital capacity (FVC) | 12 months
  Average for each study arm
Number of patients with >10% decline in FVC | 12 months
Number of patients starting new treatments for their interstitial lung disease | 12 months
Adherence to study measurements | 12 months
  Active study arm only, adherence calculated as number of days with recordings divded by 156 days, result will be an average.
Number of patients recording measurements at least once/week on at least 66% study weeks | 12 months
  active study arm only.
Number of unscheduled reviews per patient | 12 months
  Average for each study arm
Number of hospital admissions per patient | 12 months
  Average for each study arm
Change in patient recorded dyspnoea (mMRC) score | 12 months
  Average for each study arm
Change in health-related quality of life (EQ-5D-5L) score | 12 months
  Average for each study arm
Change in King's Brief Interstitial Lung Disease (K-BILD) score | 12 months
  Average for each study arm
Change in Generalised Anxiety Disorder Assessment (GAD-7) | 12 months
  Average for each study arm
Change in Patient Activation Measure (PAM-13) | 12 months
  Average for each study arm

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Wickremasinghe, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (12):
- United Kingdom (12):
  - Basingstoke and North Hampshire Hospital, Basingstoke
  - Royal Papworth Hospital, Cambridge
  - Royal Devon University Healthcare NHS Trust, Exeter
  - Leeds Teaching Hospital NHS Trust, Leeds
  - University Hospital of Leicester NHS Trust, Leicester
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Imperial College Healthcare NHS Trust, London
  - Royal Brompton Hospital, London
  - St George's University Hospital NHS Foundation Trust, London
  - Sheffield Teaching Hospitals NHS Trust, Sheffield
  - Royal Hampshire County Hospital, Winchester
  - New Cross Hospital, Royal Wolverhampton NHS Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: No
Aggregate participant data will be available to shared with other researchers only.